CLINICAL TRIAL: NCT00942812
Title: A Community Based Intervention and Evaluation of the Impact of Social Marketing of a Diarrhea Management Pack(Comprising of Low Osmolality ORS, Zinc Tablets, Water Purification Tablets and Pictorial Chart) on Childhood Diarrhea.
Brief Title: Community Based Intervention and Evaluation of the Impact of Social Marketing of a Diarrhea Management Pack
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Aga Khan University (Other)
Collaborators: John Snow, Inc. (Industry)
Responsible Party: Dr. Zulfiqar A Bhutta, Aga Khan University
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1235-Ped/ERC-09
Record Dates: First submitted 2009-07-20; First posted 2009-07-21 (Estimated); Last update posted 2011-08-10 (Estimated); Status verified 2009-07

CONDITIONS: Diarrhea
Keywords: Children; Recovery; Diarrhea Pack; Social Marketing
MeSH Terms: conditions — Diarrhea | interventions — ORALIT

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Intervention (Experimental): A diarrhea Pack comprising of low osmolality ORS, Zinc, water purification sachets and pictorial chart.
  Interventions: Other: Diarrhea Pack
- Control (Other): Standard Care through National LHW (Lady Health Workers)program
  Interventions: Other: ORS

INTERVENTIONS:
Other: Diarrhea Pack — Low osmolality ORS, Zinc tablets, water purification tablets and pictorial chart
  Arms: Intervention
Other: ORS — ORS has been supplied to diarrheal cases as standard care through the LHW program at community level
  Arms: Control

SUMMARY:
Diarrhoeal diseases are still the major paediatric health concern worldwide, contributing for 2.5 million annual deaths in children. Although the treatment of diarrhoeal illness as per the World Health Organization (WHO) guidelines brings about a considerable decline in the burden of the disease but there is still a lot to be done for this issue. Zinc supplementation along with Oral Rehydration Solution (ORS) has emerged as a potent approach to treat diarrhoea. It is believed that the children having zinc deficiency are at high risk of developing infectious diseases which eventually lead to a high burden of mortality.

In order to prevent and effectively manage diarrheal episodes, it is important that water purification tablets, zinc and oral rehydration salt is always available in each household. Though, these products are easily available in the market separately, but are rarely available together in any household. If these products are made available in a single packet, it is likely to be an effective strategy in combating diarrheal diseases in the community.

ELIGIBILITY:
Inclusion Criteria:

* Children under 5 years of age suffering from diarrhea residing in study area and having consent to participate

Exclusion Criteria:

* Failure to provide consent or children having debilitating illness or requiring emergency hospital care.

Ages: 2 Months to 59 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 7200 (Actual)
Dates: Start 2009-07; Primary Completion 2010-06 (Actual); Study Completion 2010-09 (Actual)

PRIMARY OUTCOMES:
Reduction in Diarrhea related morbidity | 1 year

CONTACTS AND LOCATIONS:
Locations (1):
- AKU Project Office, Khairpur, Sindh, Pakistan